CLINICAL TRIAL: NCT06472765
Title: Comprehensive Registry and PCR Analysis of the Vaginal Microbiome in Women: Data Collection in Healthy and Diseased States
Brief Title: Vaginal Ecosystem and Network in the United States Study
Acronym: VENUS
Status: Enrolling by invitation | Type: Observational
Sponsor: Vaginal Biome Science (Other)
Responsible Party: Sponsor
Other Study IDs: CRVA2024
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Bacterial Vaginosis; Candidiasis; Urinary Tract Infections; Genitourinary Syndrome of Menopause; Lichen Sclerosus; Lichen Planus; Vulvodynia; Endometriosis; Ureaplasma Infections; Cancer; Desquamative Inflammatory Vaginitis
MeSH Terms: conditions — Vaginosis, Bacterial; Candidiasis; Urinary Tract Infections; Lichen Sclerosus et Atrophicus; Lichen Planus; Vulvodynia; Endometriosis; Ureaplasma Infections; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Vaginal swab for Next Generation Sequencing and Polymerase Chain Reaction tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (13):
- Premenopausal Healthy: Premenopausal Healthy
  Interventions: Diagnostic Test: Vaginal Swab Collection
- Perimenopausal Healthy: Perimenopausal Healthy
  Interventions: Diagnostic Test: Vaginal Swab Collection
- Postmenopausal Healthy: Postmenopausal Healthy
  Interventions: Diagnostic Test: Vaginal Swab Collection
- Bacterial Vaginosis: Bacterial Vaginosis
  Interventions: Diagnostic Test: Vaginal Swab Collection
- Candidiasis: Yeast Infections
  Interventions: Diagnostic Test: Vaginal Swab Collection
- Urinary Tract Infection: Premenopausal and Postmenopausal Women
  Interventions: Diagnostic Test: Vaginal Swab Collection
- Genitourinary Syndrome of Menopause: Vaginal Atrophy
  Interventions: Diagnostic Test: Vaginal Swab Collection
- Lichen Sclerosus/Planus: Lichen Sclerosus/Planus
  Interventions: Diagnostic Test: Vaginal Swab Collection
- Vulvodynia: Vulvodynia
  Interventions: Diagnostic Test: Vaginal Swab Collection
- Endometriosis: Endometriosis
  Interventions: Diagnostic Test: Vaginal Swab Collection
- Ureaplasma: Ureaplasma
  Interventions: Diagnostic Test: Vaginal Swab Collection
- Desquamative Inflammatory Vaginitis (DIV): Desquamative Inflammatory Vaginitis (DIV)
  Interventions: Diagnostic Test: Vaginal Swab Collection
- Cancer: Group 1: Breast cancer patients diagnosed at stages 1-3, post-menopausal (due to surgical, chemical reasons, or age-related natural processes), and currently receiving anti-estrogen treatment for a minimum of 90 days.
  Group 2: Breast cancer patients diagnosed at stages 1-3, pre-menopausal, and undergoing anti-estrogen endocrine therapy for at least 90 days.
  Group 3: Participants diagnosed with any type of cancer at stages 1-3, not receiving anti-estrogen therapy, but have been using vaginal estrogen, prasterone, or DHEA for 90 days or more. Should not be on systemic hormone replacement therapy (estrogen with or without progesterone).
  Group 4: Diagnosed with any type of cancer at stages 1-3, and should not be receiving any anti-estrogen therapy or using vaginal estrogen, prasterone, or DHEA. These individuals must not be on systemic hormone replacement therapy.
  Group 5: Participants diagnosed at stage 4
  Interventions: Diagnostic Test: Vaginal Swab Collection

INTERVENTIONS:
Diagnostic Test: Vaginal Swab Collection — Vaginal Swab Collection

SUMMARY:
The central premise of this study is that the intricate balance and diversity of the vaginal microbiome plays a pivotal role in the onset, progression, and severity of various gynecological conditions. Specifically, the research aims to investigate how imbalances in microbial communities, such as the overgrowth of pathogenic bacteria or the depletion of beneficial ones, are linked to conditions like Bacterial Vaginosis, Candidiasis, Urinary Tract Infections, Vaginal Atrophy, and others. By employing PCR testing and the outcomes of next-generation sequencing (NGS) of the microbiome, the study seeks to identify distinct microbial profiles and patterns that are characteristic of each condition. This nuanced understanding is expected to lead to more accurate and early diagnosis, facilitating personalized and effective treatment strategies that go beyond the conventional, often indiscriminate use of antibiotics.

DETAILED DESCRIPTION:
This study protocol is developed to analyze the vaginal microbiome of women using a 56-panel PCR test and NGS test. The aim is to collect vaginal swab samples from a wide range of participants, including both healthy individuals and those with diagnosed gynecological conditions, to identify different microbiome profiles.

A key aspect of this study is the creation of a registry that will compile the data obtained from the PCR/NGS test results and participant information. This registry will serve as a valuable resource for ongoing research and will support the development of personalized approaches in women's health care. By systematically collecting and analyzing data, the registry will facilitate a better understanding of the vaginal microbiome's role in health and disease, aiding in the advancement of diagnostic and therapeutic strategies.

Additionally, the registry will provide a foundation for future studies, allowing for the exploration of long-term trends and relationships within the vaginal microbiome. This could lead to new insights into how the microbiome influences gynecological health and the development of targeted treatments. The combination of validating a precise diagnostic tool and establishing a comprehensive registry is aimed at enhancing patient care and supporting the broader research community in women's health.

ELIGIBILITY:
Inclusion Criteria:

* Healthy cis-gender women between ages 18 and 89

Exclusion Criteria:

* Pregnant or trying to conceive (i.e. IVF, IUI)

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender women
Study Population: This study's substantial sample size of 3,250 participants is statistically justified to ensure a diverse and representative sample of the population, providing increased statistical power for detecting variations in the vaginal microbiome. This approach not only allows for a comprehensive understanding of microbiome variability but also ensures the ethical utility of the research, making the findings significantly beneficial for a broad demographic. The following are the subgroups of conditions/individuals that will be sampled, each 250 swabs:
  1. Premenopausal Healthy
  2. Perimenopausal Healthy
  3. Postmenopausal Healthy
  4. Bacterial Vaginosis
  5. Candidiasis (Yeast Infections)
  6. Urinary Tract Infection (premenopausal and postmenopausal)
  7. Genitourinary Syndrome of Menopause
  8. Lichen Sclerosus/Planus
  9. Vulvodynia
  10. Endometriosis
  11. Ureaplasma
  12. Desquamative Inflammatory Vaginitis (DIV)
  13. Cancer (various types)
Sampling Method: Non-Probability Sample
Enrollment: 3250 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Microbiome Analysis | Day 1
  To analyze the vaginal microbiome in patients with diverse vaginal health conditions using next-generation sequencing (NGS) and a 56-panel PCR test to understand microbial diversity and implications for disease management.

SECONDARY OUTCOMES:
Registry | Day 1
  Data collection for future research

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Capone, PhD, Principal Investigator — Vaginal Biome Science
Locations (21):
- United States (20):
  - Women's Pelvic Health Center, Fullerton, California
  - Claris Health, Los Angeles, California
  - University of California Los Angeles Department of Radiation Oncology, Los Angeles, California
  - Pelvic Pain Rehab, Pasadena, California
  - Healthy Mothers, Healthy Babies Coalition of Hawaii, Honolulu, Hawaii
  - Rachel Rubin MD PLLC, Bethesda, Maryland
  - Dr. Christina Enzmann at Easton Advanced Aesthetics and Regenerative Medicine, Easton, Maryland
  - Empowered Midwifery and Wellness LLC, Alexandria, Minnesota
  - Xena Health, Henderson, Nevada
  - Empire OBGYN, Kenmore, New York
  - Gary H Goldman, MD, New York, New York
  - Camel City Women's Wellness, Winston-Salem, North Carolina
  - UH Hospitals, Mayfield Heights, Ohio
  - Northwest Obstetrics and Gynecology, Oklahoma City, Oklahoma
  - Haven Center for Sexual Medicine & Vulvovaginal Disorders, Tulsa, Oklahoma
  - Center of the Health, Corvallis, Oregon
  - Amber Wellness Group, Portland, Oregon
  - Center for Pelvic Medicine, Bryn Mawr, Pennsylvania
  - North Houston Gynecologic Oncology Surgeons, PLLC, Shenandoah, Texas
  - Hello Climax, Virginia Beach, Virginia
- Integrative Naturopathic Medical Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided